CLINICAL TRIAL: NCT03212911
Title: Immunogenicity and Safety of 4- vs. 3-standard Doses HBV Vaccination in HIV-infected Adults With Isolated Anti-HBc Antibody
Brief Title: HBV Vaccination in HIV-infected Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04565
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis B Vaccination, HIV
Keywords: HBV vaccination, HIV, isolated anti-HBc
MeSH Terms: interventions — Hepatitis B Vaccines

STUDY DESIGN:
Intervention Model Description: Open-label, randomized controlled trial (RCT) with 1:1 allocation in parallel arms
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-standard dose HBV vaccination group (Active Comparator): participants will receive 3 standard doses of HBV vaccination at 0, 1, 6 months
  Interventions: Biological: Hepatitis B vaccine
- 4-standard dose HBV vaccination group (Active Comparator): participants will receive 4 standard doses of HBV vaccination at 0, 1, 2, 6 months
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Hepatitis B vaccine — Hepatitis B vaccine (20 mcg/ml) 1 ml intramuscular injection in 3 (at 0, 1, 6 months) or 4 doses (0, 1, 2, 6 months)

SUMMARY:
The finding of isolated hepatitis B core antibody (isolated HBc) in absent of recent active hepatitis could cause by several scenarios, including false positive, remote infection without viremia, and occult infection with low viremia. Hepatitis B virus (HBV) vaccine booster could be a great prevention strategy for those who do not have HBV viremia. There is no standard consensus for management of this issue especially among HIV infected population. In addition, prior studies revealed that HIV-infected individuals had lower immunologic response to HBV vaccine than general population. This study intends to compare the immune response and safety of 4- versus 3-standard dose of hepatitis B virus vaccination in HIV-infected adults who has isolated HBc. The immunologic response will be evaluated after the participants receive vaccination.

DETAILED DESCRIPTION:
* A randomized controlled trial to evaluate differences in immunogenicity and safety of the two hepatitis B vaccination regimens, including the percentage of responders, high-level responders, anamnestic response, geometric mean titers of anti-HBs antibody, adverse events and predictive factors associated with vaccine responsiveness
* After participant enrollment, data on baseline characteristics, time since HIV diagnosis, CD4 counts, HIV viral load, antiretroviral treatment regimen and duration will be collected, then the participants will be randomized into 2 groups to receive either 3- or 4-standard doses (20 mcg per dose) of HBV vaccination, and follow-up blood test for anti-HBs titers at multiple pre-specified time points to evaluate outcomes

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* On combination antiretroviral therapy (cART)
* CD4 ≥ 200 cell/mm3 for ≥ 1 year
* HIV viral load < 20 copies/ml for ≥ 1 year
* Isolated anti-HBc Ab (negative HBsAg, anti-HBs Ab) and negative anti-HCV at screening

Exclusion Criteria:

* Pregnancy
* Previous HBV vaccination
* Intolerance to any component of HBV vaccine
* Transaminitis in the past 3 months (≥ 5 UNL)
* Ongoing opportunistic infection (OI)
* Active malignancy, with current chemotherapy or radiotherapy
* Systemic steroid therapy (≥ 0.5 mg/kg/day) or any immunomodulating therapy in the last 6 months
* Other immunocompromised disorders (e.g. solid organ transplant)
* Asplenism
* Renal insufficiency (CrCl ≤ 30 mL/min)
* Decompensated cirrhosis (Child-Pugh C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Immunologic response to 4 versus 3 doses of HBV vaccination in HIV-infected adults with isolated anti-HBc antibody, demonstrated by percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL ) at week 28 | 28 weeks after the first dose of HBV vaccination
  Immunologic response to 4 versus 3 doses of HBV vaccination in HIV-infected adults with isolated anti-HBc antibody, demonstrated by percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL ) at week 28

SECONDARY OUTCOMES:
Anamnestic response at week 4 | 4 weeks after the first dose of HBV vaccination
  Anamnestic response at week 4
Percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL) at month 12 | 12 months after the first dose of HBV vaccination
  Percentage of responders (with anti-HBs Ab ≥ 10 mIU/mL) at month 12
Percentage of high-level responders (with anti-HBs Ab ≥ 100 mIU/mL) at week 28 and month 12 | 28 weeks and 12 months after the first dose of HBV vaccination
  Percentage of high-level responders (with anti-HBs Ab ≥ 100 mIU/mL) at week 28 and month 12
Intensity and frequency of vaccine adverse event (AE) | 1 year
  Intensity and frequency of vaccine adverse event (AE)
Geometric mean titers of anti-HBs Ab at week 28 and month 12 | 28 weeks and 12 months after the first dose of HBV vaccination
  Geometric mean titers of anti-HBs Ab at week 28 and month 12
Predictive factors associated with response to vaccine (age, sex, CD4 count) | 1 year
  Predictive factors associated with response to vaccine (age, sex, CD4 count)

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of medicine, Chiang Mai University, Muang, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laksananun N, Praparattanapan J, Kotarathititum W, Supparatpinyo K, Chaiwarith R. Immunogenicity and safety of 4 vs. 3 standard doses of HBV vaccination in HIV-infected adults with isolated anti-HBc antibody. AIDS Res Ther. 2019 May 3;16(1):10. doi: 10.1186/s12981-019-0225-3. PMID 31053142